CLINICAL TRIAL: NCT04443049
Title: To Study the Effects of Addition of Mebendazole to Lenvatinib in Cirrhotics With Advanced Hepatocellular Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-32
Record Dates: First submitted 2020-06-15; First posted 2020-06-23 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — lenvatinib; Mebendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib +Placebo (Active Comparator): Lenvatinib will be given once a day(OD) orally at dose of 8 mg if body weight is < 60 kg and 12 mg if body weight is > 60 kg ) with placebo (Tab Mecovit) orally twice a day (BD) daily
  Interventions: Drug: Lenvatinib; Other: Placebo
- Lenvatinib and mebendazole (Experimental): Lenvatinib will be given orally once a day (OD) at dose of 8 mg if body weight is < 60 kg and 12 mg if body weight is > 60 kg) and mebendazole will be given at dose of 100 mg orally twice a day (BD) daily
  Interventions: Drug: Lenvatinib; Drug: Mebendazole

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be given once a day(OD) orally at dose of 8 mg if body weight is < 60 kg and 12 mg if body weight is > 60 kg
Drug: Mebendazole — mebendazole will be given at dose of 100 mg orally twice a day (BD) daily
  Arms: Lenvatinib and mebendazole
Other: Placebo — Placebo (Tab Mecovit) orally twice a day (BD) daily
  Arms: Lenvatinib +Placebo

SUMMARY:
Currently the available first line palliative therapy for advanced HCC is Sorafenib and Lenvatinib of which Lenvatinib is tolerated better. Unfortunately, patients tend to progress after few months of therapy. Therefore it is imperative, to do trials by combinative therapy to the available therapy for added survival benefits and quality of life with advanced HCC. In this regard, Mebendazole appears to be a good choice for drug repurposing as it has shown very promising results either alone or in combination with other therapies in tumors of GI origin and CNS tumors. With regard to HCC Mebendazole has been found to be effective in vitro system of HCC and preclinical models. However no clinical trials have been initiated till now. The key hallmark features of HCC include activation of MAPK and angiogenesis which in turn are targeted by RTK inhibitors such as Sorafenib and Lenvatinib. In this regard Mebendazole has broad range of action by not only inhibiting angiogenesis and pro-survival pathways of MAPK, but by also inhibiting the secretion of MMPs and Tubulin polymerization which can all be beneficial in tumor regression and prevention of chemo-resistance in HCC. Mounting of a strong immune response plays an important role in identification of tumor antigen and thereby clearing of tumors. While Mebendazole can modulate the tumor, the data is scant with respect to the role of the drug. Hence repurposing Mebendazole as a combinatorial therapy appears a promising approach and forms the basis of the present work. We hypothesize that combinatorial therapy of addition of mebendazole to lenvatinib will prove more beneficial than lenvatinib alone in increasing the overall survival of patients with advanced HCC. To prove the mechanistic effects of mebendazole on HCC, we will also conduct a animal study in preclinical mice model of HCC with the help of our animal house facility. The animal study will help us to understand the additional benefits from mebendazole and lenvatinib with objective evidence of liver biopsy which is not feasible in humans.

DETAILED DESCRIPTION:
(A) STUDY HYPOTHESIS

* Mebendazole augments response of lenvatinib by synergistic response.
* Addition of anti angiogenic drugs (lenvatinib and mebendazole) to hypoxic environment generated post locoregional therapy like TACE leads to more effective control of advanced HCC resulting in improvement in overall survival.

(B) AIM: To compare the efficacy of combination of mebendazole with lenvatinib in cirrhotics with advanced Hepatocellular Carcinoma.

(C) OBJECTIVE:

Primary objective:

To compare the efficacy of combination of mebendazole with lenvatinib in improving the overall survival at 15 months in cirrhotics with advanced HCC.

Secondary objective:

1. To compare the progression free survival with combination therapy of mebendazole and lenvatinib in advanced Hepatocellular Carcinoma (HCC).
2. To compare the objective response rate (ORR), disease control rate (DCR) and clinical benefit rate (CBR) with combinative therapy of mebendazole and lenvatinib in advanced HCC.
3. To study therapy related adverse effects of mebendazole in cirrhotics.
4. To develop pre-clinical HCC animal model to prove the added efficacy of combination therapy.

(D)STUDY DESIGN Type of study - Single center, prospective, open label, randomized control study Study population - cirrhosis of liver of any etiology with advanced HCC undergoing at ILBS Study duration - 22 months from the date of approval of IEC Sample size - Considering mebendazole adds 2 months more to lenvatinib which offers 13 months overall survival, power of the study as 80 %, attrition rate as 30 %, alpha error of 5%, sample size will be 85 patients in each arm ( totally 170 patients).

(F) Methodology: Cirrhotics with advanced HCC proven by imaging and or biopsy or cytology, fulfilling the eligibility criteria will be enrolled in the study. They may undergo 1 or 2 sessions of locoregional therapy (TACE/ SBRT/RFA) if feasible. All patients will undergo complete physical examination, CBC, LFT, KFT, INR, AFP, PIVKAII, CEMRI/ CECT upper abdomen (Triple phase ), UGI endoscopy at baseline before randomization.

Randomization:

Those patients who are not feasible for locoregional therapy will be randomized at baseline. Those patients undergoing locoregional therapy will be randomized after 1 month of last locoregional therapy (patient may undergo maximum of two sessions of locoregional therapy before randomization). The response will be determined by m RECIST criteria before randomization. Those patients requiring further sessions of locoregional therapy beyond two sessions will not be randomized into study.

Patient will be then randomized to one of the two groups Arm I :Lenvatinib +Placebo( Lenvatinib will be given once a day(OD) orally at dose of 8 mg if body weight is < 60 kg and 12 mg if body weight is > 60 kg ) with placebo (Tab Mecovit) orally twice a day (BD) daily Arm II : Lenvatinib and mebendazole ( Lenvatinib will be given orally once a day (OD) at dose of 8 mg if body weight is < 60 kg and 12 mg if body weight is > 60 kg) and mebendazole will be given at dose of 100 mg orally twice a day (BD) daily

Follow-up Patients will be followed up with clinical events, CBC, LFT, KFT, INR, AFP, PIVKAII, CEMRI/ CECT upper abdomen (Triple phase ) at the end of 1 month, 3 months, 6 months, 9 months, 12 months and 15 months.

INVESTIGATIONS AND FOLLOW UP At Baseline (before therapy) and during follow up

* Hematology- repeated at the end of 1, 3, 6, 9, 12, 15 months.

  - CBC
* Biochemistry - repeated at the end of 1, 3, 6, 9, 12, 15 months.

  * Serum Electrolytes, Kidney function test
  * Liver function test, INR
* CTP and MELD scores
* AFP, PIVKA II - repeated at the end of 1, 3, 6, 9, 12, 15 months.
* UGIE at baseline
* CEMRI / CECT upper abdomen - Triple phase - repeated at the end of 1, 3, 6, 9, 12, 15 months.
* PET CT - if systemic spread suspected or else at the end of 6 and 15 months
* Liver Biopsy/FNAC will be done in cases where its clinically indicated.

The pre-clinical model will be developed in mice, for which separate application will be submitted to the animal ethics committee of the institute.

Timeline of follow up

* At the end of first month
* Then every 3 months until 15 months after starting therapy

STATISTICAL ANALYSIS

* Data will be reported as mean + SD
* Categorical variables will be compared using the chi-square test or Fisher exact test
* Normal continuous variables will be compared using the Student t test
* Non normal continuous variables will be compared using the Mann-Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data).
* Comparison between groups on quantitative variables will be analyzed by ANOVA
* The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test
* A Cox regression analysis will be performed to identify independent prognostic factors for survival.

Intervention: This Randomized Controlled trial will be conducted at Institute of Liver & Biliary SciencesLBS New Delhi between June 2020 and March 2022

Salvage therapy

* TACE or TARE if progressive disease
* Nivolilumab if the patient had a progressive disease at 6 months of therapy

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of Liver with HCC on imaging and/or biopsy or cytology
* Child Pugh A, Child Pugh B < 8
* Advanced HCC - as defined by BCLC - C
* ECOG Performance Status 1-2
* Adequately controlled blood pressure (BP) with up to 3 antihypertensive agents, defined as BP ≤150/90 millimeters of mercury (mmHg) at screening and no change in antihypertensive therapy within 1 week prior to commencement of intervention.
* Valid Consent
* Age 18-70 years

Exclusion Criteria:

* Decompensated Cirrhosis
* Child Pugh C, Child Pugh B > 7
* HCC patients with a curative therapy (RFA/MWA or LT)
* Prior systemic therapies (or) immunotherapy for HCC
* ECOG Performance Status 3-4
* Post Liver transplant HCC recurrence
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-06-19 (Estimated); Study Completion 2022-06-19 (Estimated)

PRIMARY OUTCOMES:
Overall survival in both groups | 15 months
Death | 2 year
Progressive disease requiring change of therapy in both groups | 2 year

SECONDARY OUTCOMES:
Progressive disease requiring quitting therapy in both groups | 2 year
Therapy related adverse effects in both groups | 2 year
Worsening of performance status in both groups | 2 year
  Worsening of performance will be measured by Eastern Cooperative Oncology Group (ECOG) Criteria.
Decompensation of underlying cirrhosis in both groups | 2 year
  Barcelona-Clinic Liver Cancer (BCLC) staging classification will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided